CLINICAL TRIAL: NCT00188240
Title: Insulin Resistance Associated With Chronic Hepatitis C (CHC) and the Effect of Anti-Viral Therapy
Brief Title: Insulin Resistance Associated With Chronic Hepatitis C (CHC) and the Effect of Antiviral Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03-0510-AE 04-0292-A
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2005-11-29 (Estimated); Status verified 2005-09

CONDITIONS: Hepatitis C; Hepatitis B
Keywords: hepatitis C; insulin resistance; antiviral therapy
MeSH Terms: conditions — Hepatitis C; Hepatitis B; Insulin Resistance | interventions — peginterferon alfa-2a; Ribavirin

INTERVENTIONS:
Drug: Pegasys; Copegus.

SUMMARY:
The literature suggests that there may be an association between hepatitis C and type 2 diabetes mellitus independent of the presence of cirrhosis, the likely mechanism for which is insulin resistance. The prevalence of insulin resistance in patients with hepatitis C is unknown. Furthermore, there are no studies that indicate an increased prevalence of insulin resistance in patients with hepatitis C compared to other etiologies of liver disease. The role that hepatitis C may have in the development of insulin resistance is unclear. The effect of antiviral therapy for hepatitis C virus on insulin resistance has not been addressed. The long-term consequence of insulin resistance is type 2 diabetes mellitus. There is significant morbidity and mortality from type 2 diabetes mellitus in the general population, and similar complications would be expected in patients with hepatitis C and insulin resistance particularly if they develop type 2 diabetes mellitus.

Our hypothesis: The prevalence of insulin resistance is increased in patients with chronic hepatitis C compared to chronic hepatitis B. Secondarily, insulin resistance when present in patients with chronic hepatitis C improves with successful antiviral therapy.

This study has two phases. The first phase of our study will be to estimate the prevalence of insulin resistance in individuals with chronic hepatitis C without cirrhosis compared to patients with chronic hepatitis B without cirrhosis. The second phase of the study will be restricted to those patients with hepatitis C found to be insulin resistant from phase 1, in the absence of known risk factors for insulin resistance (cirrhosis, diabetes). The effect on insulin resistance of anti-viral therapy to eradicate hepatitis C will be assessed.

DETAILED DESCRIPTION:
The first phase will include patients with hepatitis C who are candidates for anti-viral treatment, and patients with chronic hepatitis B who have undergone a recent liver biopsy showing hepatitis without cirrhosis, with equal numbers in each group (100/ group).

Phase 2 (40 patients)- Patients with hepatitis C found in phase 1 by the HOMA test to have increased insulin resistance will be recruited to phase 2 (interventional phase). Patients with HBV infection will not be studied further.

The study will be conducted at a single center using an open-label design. All patients will be treatment naïve. Up to 40 patients will be treated per current standard of care with combination pegylated interferon alfa and ribavirin (Phase 2). Patients with genotype 2 or 3 will be treated with combination weekly Pegasys with a daily Copegus dose of 800 mg given for 24 weeks (Group A). Patients with genotype non-2 or 3 will be treated with combination weekly Pegasys with a daily Copegus dose of 1000-1200 mg given for 48 weeks (Group B). Both groups will have an untreated follow-up period of 24 weeks. Pegasys will be administered sc once weekly (180 microg in 0.5 or 1 mL solution) and Copegus will be taken po daily in split doses of 400 mg in the morning and 400 mg in the evening (i.e., 2 tablets of 200 mg bid). For doses of 1000 mg (genotype non- 2 or 3 patients whose body weight < 75 kg) Copegus will be administered po daily: 400 mg (i.e. 2 tablets of 200 mg) in the morning and 600 mg (i.e. 3 tablets of 200 mg) in the evening. For genotype non-2 or 3 patients whose body weight is 75 kg, 600 mg (i.e. 3 tablets of 200 mg) in the morning and 600 mg (i.e. 3 tablets of 200 mg) in the evening is recommended. All patients in this study will receive Copegus treatment with food. By definition, Copegus "with food" means taking their doses within 1 hour before or 2 hours after a meal. The meal should be considered "regular" as opposed to "fat-restricted".

All 40 patients who meet inclusion criteria will also have indices of body fat assessed through calculation of their BMI, DEXA scanning, and waist-to-hip circumference measurements. Prior to therapy all patients will undergo the OGTT , which is a dynamic test for insulin resistance providing accurate information on the relationship between insulin and glucose.

At week 12 of treatment patients will have a quantitative assessment of HCV viral load and a second OGTT . The current standard of therapy is to discontinue anti-viral therapy in patients with genotype 1 or 4 without a ≥ 2-log fall in HCV RNA. Those who have a ≥ 2-log fall in HCV RNA are expected to have a SVR. Patients to be continued on anti-viral therapy will then be followed to SVR.

Twenty-four weeks after completion of anti-viral therapy, a OGTT will be repeated (SVR OGTT). The effect of viral clearance on insulin resistance will be assessed by comparing the OGTT at SVR (SVR OGTT) to pre-treatment OGTT.

Patients who are Non-Responders should also be assessed for safety 4-8 weeks after their last dose of test medication following premature discontinuation from the study. Non-Responders are defined as patients without a 2-log drop in PCR between baseline and week 12 or a positive PCR at their last visit. Responders should be followed for until Week 48 (Group A patients) or Week 72 (Group B patients). Responders are defined as patients who have a 2-log drop in PCR between baseline and week 12 and a negative PCR at their last visit. Female patients receiving Copegus should continue to do the home-based pregnancy test every 4 weeks for the 6-month period after the last dose of study drug.

Efficacy assessments consist of serum HCV-RNA via PCR. Quantitative viral titers (AMPLICOR HCV MONITOR Test, v2.0) will be obtained at Weeks 0 and 12 from all patients. Qualitative HCV-RNA results (AMPLICORÒ HCV Test, v2.0) will be obtained at treatment period Week 24 for all patients and Week 48 for group B; in addition during follow-up at week 24 for all patients.

Insulin resistance as determined by the OGTT method will be assessed prior to initiation of therapy, at 12 weeks of therapy, and during follow-up at week 24 for all patients.

Study Outcome:

Phase 1 - To evaluate the prevalence of insulin resistance in patients with hepatitis C without cirrhosis and compare it to that observed in patients with hepatitis B also without cirrhosis.

Phase 2 - Interventional phase - To evaluate the effect of anti-viral therapy on insulin resistance, determined by the OGTT method, in patients with hepatitis C found to have insulin resistance pre-treatment.

- To evaluate the safety, efficacy and tolerability of Pegasys (peginterferon alfa-2a) given in combination with Copegus (ribavirin) given for 24 weeks or 48 weeks in treatment naïve patients with chronic hepatitis C (CHC).

ELIGIBILITY:
Inclusion Criteria:

* patients attending Liver Clinic at Toronto Western Hospital, Toronto, ON, Canada
* Male and female patients
* Serologic evidence of chronic hepatitis C infection by an anti-HCV antibody test
* Detectable serum HCV-RNA
* Negative urine or blood pregnancy test (for women of childbearing potential) documented within the 24-hour period prior to the first dose of study drug
* All fertile males and females receiving Copegus must be using two forms of effective contraception during treatment and during the 6 months after treatment end
* All patients should have insulin resistance (>2.1) determined by the homeostasis model assessment (HOMA) method.

Exclusion Criteria:

* Women with ongoing pregnancy or breast feeding
* Therapy with any systemic anti-neoplastic or immunomodulatory treatment (including supraphysiologic doses of steroids and radiation) < 6 months prior to the first dose of study drug
* Any investigational drug < 6 weeks prior to the first dose of study drug
* Co-infection with active hepatitis A, hepatitis B and/or human immunodeficiency virus (HIV)
* History or other evidence of a medical condition associated with chronic liver disease other than HCV (e.g., hemochromatosis, autoimmune hepatitis, metabolic liver disease, alcoholic liver disease, toxin exposures)
* Signs or symptoms of hepatocellular carcinoma
* History or other evidence of bleeding from esophageal varices or other conditions consistent with decompensated liver disease
* Neutrophil count <1500 cells/mm3 or platelet count <90,000 cells/mm3 at screening
* Serum creatinine level >1.5 times the upper limit of normal at screening
* History of severe psychiatric disease, especially depression. Severe psychiatric disease is defined as treatment with an antidepressant medication or a major tranquilizer at therapeutic doses for major depression or psychosis, respectively, for at least 3 months at any previous time or any history of the following: a suicidal attempt, hospitalization for psychiatric disease, or a period of disability due to a psychiatric disease
* History of a severe seizure disorder or current anticonvulsant use
* History of immunologically mediated disease, chronic pulmonary disease associated with functional limitation, severe cardiac disease, major organ transplantation or other evidence of severe illness, malignancy, or any other conditions which would make the patient, in the opinion of the investigator, unsuitable for the study
* History of thyroid disease poorly controlled on prescribed medications, elevated thyroid stimulating hormone (TSH) concentrations with elevation of antibodies to thyroid peroxidase and any clinical manifestations of thyroid disease
* Evidence of severe retinopathy (e.g. CMV retinitis, macula degeneration)
* Evidence of drug abuse (including excessive alcohol consumption) within one year of study entry
* Inability or unwillingness to provide informed consent or abide by the requirements of the study
* Cirrhosis on liver biopsy
* Type II diabetes mellitus
* Diabetogenic medications including steroids
* Current daily alcohol use of greater than 20 gm
* Known hypersensitivity to any of the contents of the study drug
* Patients currently participating in other Clinical Trials
* Patients previously treated for hepatitis C / received alfa-interferon

Additional exclusion criteria for patients receiving Copegus:

* Male partners of women who are pregnant
* Hgb <12 g/dL in women or <13 g/dL in men at screening
* Any patient with an increased baseline risk for anemia (e.g. thalassemia, spherocytosis, history of GI bleeding, etc) or for whom anemia would be medically problematic
* Patients with documented or presumed coronary artery disease or cerebrovascular disease should not be enrolled if, in the judgment of the investigator, an acute decrease in hemoglobin by up to 4 g/dL (as may be seen with Copegus therapy) would not be well-tolerated

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2003-08

PRIMARY OUTCOMES:
Phase I - To evaluate the prevalence of insulin resistance in patients with hepatitis C without cirrhosis and compare it to that observed in patients with hepatitis B also without cirrhosis.
Phase II - Interventional phase - To evaluate the effect of anti-viral therapy on insulin resistance, determined by the OGTT method, in patients with hepatitis C found to have insulin resistance pre-treatment.
- To evaluate the safety, efficacy and tolerability of Pegasys (peginterferon alfa-2a) given in combination with Copegus (ribavirin) given for 24 weeks or 48 weeks in treatment naïve patients with chronic hepatitis C (CHC).

CONTACTS AND LOCATIONS:
Overall Officials: E.J.L (Jenny) Heathcote, MD, Principal Investigator — UHN - Toronto Western Hospital, University of Toronto
Locations (1):
- Liver Clinic, Toronto Western Hospital, UHN., Toronto, Ontario, Canada